CLINICAL TRIAL: NCT05709132
Title: Implementation and Preliminary Effectiveness Evaluation of the iPeer2Peer Support Mentorship Program for Adolescent and Transitioning Heart Function Patients
Brief Title: iP2P Mentorship Program for Adolescent HF Patients
Acronym: iP2P HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Centre Hospitalier Universitaire Sainte-Justine (Unknown); University of Alberta/Stollery Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Samantha Anthony, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000080204
Record Dates: First submitted 2023-01-24; First posted 2023-02-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: Peer Support Mentorship; Pediatrics; Adherence; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: Quasi-experimental single arm pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- iPeer2Peer Program (Experimental): Participates in the iPeer2Peer program
  Interventions: Behavioral: iPeer2Peer Program

INTERVENTIONS:
Behavioral: iPeer2Peer Program — Behavioral: iPeer2Peer Support Mentorship Program is an online peer support mentorship program that has been established in multiple chronic disease populations as a self-management intervention, including chronic pain and juvenile idiopathic arthritis. The iPeer2Peer program provides modeling and reinforcement by pre-screened and trained young adult peer mentors to adolescent mentees.

SUMMARY:
The iPeer2Peer (iP2P) program is an online peer support mentorship program that provides modelling and reinforcement by trained young adult peer mentors to adolescent mentees with the same condition. A quasi-experimental single-arm pre-post study design will be employed across three sites. We will recruit 40 mentees (12-17 years of age) and 12-15 mentors (18-30 years of age) who will undergo training in mentoring and the use of eHealth technology. Mentor-mentee pairings will connect over 15 weeks through video calls and text messaging to provide peer support and encourage disease self-management skills. Data will be collected using standardized instruments and interviews across three time points.

ELIGIBILITY:
Mentee inclusion criteria:

1. patient with a cardiac diagnosis,
2. at least 4 months post-diagnosis,
3. between the ages of 12 and 17 years,
4. able to speak and read English, and
5. willingness to commit to 5-10 texts and/or calls of 20-30 minutes each with a peer mentor over a period of 15 weeks.

Mentor inclusion criteria:

1. patient with a cardiac diagnosis,
2. between the ages of 18 and 30 years,
3. able to speak and read English,
4. nominated by a member of their health care team as a good mentor based on maturity and emotional stability,
5. willingness to commit to peer mentor training (20 hours) via the PHIPA-compliant version of Zoom or Microsoft Teams and mentoring adolescent participants (once paired with mentee, 5-10 texts and/or calls of 20-30 minutes over a period of 15 weeks),
6. good communication skills (as assessed by a healthcare provider), and
7. previous experience in a professional environment (e.g., as a camp counsellor, part time job, volunteering) is an asset.

Exclusion Criteria:

1. significant cognitive impairments as assessed by a qualified healthcare provider,
2. a diagnosis of an active psychological disorder (e.g., Major Depressive Disorder, Generalized Anxiety Disorder) likely to influence assessment of health-related quality of life and/or interfere with their ability to manage their heart failure care regimen (a diagnosis of an active psychological disorder will be determined for mentees through medical chart review and self-reported by mentors), and
3. participating in other peer support or self-management interventions.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-04-13 (Estimated); Study Completion 2027-04-13 (Estimated)

PRIMARY OUTCOMES:
Acceptability (Mentees) | 15 weeks after baseline/immediately after the intervention
  Whether the innovation is agreeable, palatable or satisfactory
Acceptability (Mentors) | Study completion, an average of 1 year
  Whether the innovation is agreeable, palatable or satisfactory
Adoption (Mentees) | Baseline to 12 weeks post-program completion
  The intention, initial decision or action to try or use an innovation
Adoption (Mentors) | Baseline to study completion, an average of 1 year
  The intention, initial decision or action to try or use an innovation
Feasibility (Mentees) | Baseline to 12 weeks post-program completion
  The extent to which an innovation can be used or carried out successfully in a given setting
Feasibility (Mentors) | Baseline to study completion, an average of 1 year
  The extent to which an innovation can be used or carried out successfully in a given setting
Appropriateness (Mentees) | Baseline to 12 weeks post-program completion
  The perceived fit, relevance or compatibility of the innovation for a practice setting; and/or its perceived fit to address an issue or problem
Appropriateness (Mentors) | Baseline to study completion, an average of 1 year
  The perceived fit, relevance or compatibility of the innovation for a practice setting; and/or its perceived fit to address an issue or problem
Level of engagement (Mentees) | 15 weeks after baseline/immediately after the intervention
Level of engagement (Mentors) | Study completion, an average of 1 year

SECONDARY OUTCOMES:
Disease self-management skills (Mentees) | Baseline to 12 weeks post-program completion
Adherence (Mentees) | Baseline to 12 weeks post-program completion
  Clinic attendance, completion of scheduled tests and procedures, and adolescent medication barriers scale
Quality of life (Mentees) | Baseline to 12 weeks post-program completion
Perceived social support (Mentees) | Baseline to 12 weeks post-program completion
Emotional distress (Mentees) | Baseline to 12 weeks post-program completion
Resiliency (Mentees) | Baseline to 12 weeks post-program completion
Assessment of mentor quality (Mentees) | 15 weeks after baseline/immediately after the intervention
Physical and emotional symptoms (Mentors) | Baseline to study completion, an average of 1 year
Perceived social role satisfaction (Mentors) | Baseline to study completion, an average of 1 year
Self-efficacy (Mentors) | Baseline to study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Anthony, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No